CLINICAL TRIAL: NCT04327076
Title: Clinical Application of Magnetically Guided Endotracheal Intubation and Airway Cleaning Robot System
Brief Title: Magnetically Guided Endotracheal Intubation and Airway Cleaning Robot System
Acronym: MGEIAACRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: XJTU1AF2015LSL-046-1
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: General Anesthesia
Keywords: Endotracheal intubation; Airway cleaning

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Robot system intervention (Experimental): 1. Evaluate the patient and sign the informed consent
  2. The patient was given general anesthesia
  3. Use magnetically guided tracheal intubation and airway cleaning robot system
  Interventions: Device: Using robot system of endotracheal intubation and airway cleaning

INTERVENTIONS:
Device: Using robot system of endotracheal intubation and airway cleaning — 1. Using the control screen to control the machine, the device first extends the intubation guide rail to the mouth of the patient's oropharyngeal ventilation tube, first sends the magnetic guide strip into the epigarynx, and at the same time, extends the magnetic anchoring unit to the patient's neck. The external magnetic anchoring unit can sense and attract the magnet on the magnetic guide strip. At this point, the machine can send the guide strip into the respiratory tract.
  2. Then, the control machine sends the tracheal intubation into the airway along the guide strip, and completes the balloon inflation to complete the endotracheal intubation operation.
  3. During or after the operation, when the sputum suction operation is needed, the parameters of the sputum suction machine are set on the operation screen to start the sputum suction operation, and the suction robot completes the sputum suction operation automatically.

SUMMARY:
Endotracheal intubation refers to the use of special equipment, through the nasal cavity or oral cavity, through the throat, glottis, the process of inserting the endotracheal tube into the trachea or bronchus. Its main function is to maintain respiratory tract patency, positive pressure ventilation and removal of respiratory secretions. Endotracheal intubation and sputum suction are important parts of first aid and surgical anesthesia. Our team developed a magnetic navigation tracheal intubation and airway cleaning robot system to achieve mechanization and integration of surgical anesthesia, airway management. This study is designed to investigate the safety and efficacy of the Magnetic navigation tracheal intubation and airway cleaning robot.

DETAILED DESCRIPTION:
Endotracheal intubation is a highly professional technique, especially for emergency patients with shallow coma, closed teeth and awake, it is more difficult to intubate. If the operation is improper, it is easy to damage the wound, pharynx and teeth or stimulate the throat to produce choking, breath holding, laryngospasm, aggravating hypoxia and mucosal injury. At present, the data of endotracheal intubation show that even under the non-emergency state of routine operation, the success rate of the first endotracheal intubation is 70%, and the success rate of secondary intubation is 89%. Under the pre-hospital emergency, the success rate of first intubation of ambulancemen is less than 50%, which is much lower than that of professional physicians. Therefore, it is of great significance to simplify the labor intensity of anesthesiologists and improve the intelligence of clinical operation.

In this study, the electromagnetic acousto-optic fusion navigation technology is used to make a half-helmet type multi-axis magnetic coupling driving navigation robot cover on the left side of the patient's head in the supine position, automatically feeding the guide core with the internal magnetic tip through the external guide tube and intubating the trachea to the pharynx, applying the attraction of the external magnet to the neck hyoid so that the magnetic tip of the guide core in the endotracheal intubation points to the glottis. With the help of internal and external magnetic attraction and moderate driving force to push the guide core into the tube first, electromagnetic induction detection and spot image analysis determine it, continue to use the magnetic coupling device to push the guide bar to the bifurcation protuberance of the trachea, fix the guide bar, push the trachea intubation to the appropriate position, and then exit the guide bar and inflate the balloon.

Sputum suction robot that can perform the sputum suction of a nurse simply, safely and effectively. It can be equipped with a closed sputum suction tube commonly used in clinical practice for sputum suction. And through a wired connection, the operator can perform sputum suction through the control unit at a long distance. In order to ensure that the machine is suitable for different patients and to ensure the safety of use, our equipment can set different depths of tube inlet, tube inlet speed, tube withdrawal speed, and sputum suction mode, while the sputum suction robot performs the entire process of sputum suction In this case, there is no need to stop the oxygen supply to the patient, and the risk of iatrogenic damage to the patient by hypoxia is also reduced To realize the mechanization and integration of surgical anesthesia and airway management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients about to undergo general anesthesia.
2. Age >18 years.
3. Informed consent obtained.
4. Generally in good condition before operation.

Exclusion Criteria:

1. Patients are unwilling to this procedure.
2. Patients with Patient has maxillofacial mass, oropharyngeal mass, neck mass.
3. Patients with loose teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-08-05 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
success rate of endotracheal intubation | measured at the time of the end of endotracheal intubation，up to 1 hour
  Success rate of single endotracheal intubation by using robot system
success rate of airway cleaning | measured at the time of the end of airway cleaning，up to 1 hour
  The success rate of airway cleaning by using robot system

SECONDARY OUTCOMES:
complications of endotracheal intubation and airway cleaning robot system | measured at the time of the end of endotracheal intubation and airway cleaning robot system,up to 1 week
  the complications of endotracheal intubation and airway cleaning robot system,including mistakenly inserted into the esophagus,teeth loose or fall out,Laryngeal edema,respiratory cardiac arrest,poorly ventilated,atelectasis,Tracheoesophageal fistula,tracheal mucosal injury,bleeding,etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lv, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Qiang Wang, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Mwakanyanga ET, Masika GM, Tarimo EAM. Intensive care nurses' knowledge and practice on endotracheal suctioning of the intubated patient: A quantitative cross-sectional observational study. PLoS One. 2018 Aug 16;13(8):e0201743. doi: 10.1371/journal.pone.0201743. eCollection 2018. PMID 30114257
- [Background] Stewart MG. Classics from The Laryngoscope: Celebrating 120 years of impact. Laryngoscope. 2015 Oct;125(10):2237. doi: 10.1002/lary.25271. Epub 2015 Sep 5. No abstract available. PMID 26341863
- [Background] Xu Z, Ma W, Hester DL, Jiang Y. Anticipated and unanticipated difficult airway management. Curr Opin Anaesthesiol. 2018 Feb;31(1):96-103. doi: 10.1097/ACO.0000000000000540. PMID 29176376
- [Background] Hsu HT, Chou SH, Wu PJ, Tseng KY, Kuo YW, Chou CY, Cheng KI. Comparison of the GlideScope(R) videolaryngoscope and the Macintosh laryngoscope for double-lumen tube intubation. Anaesthesia. 2012 Apr;67(4):411-5. doi: 10.1111/j.1365-2044.2011.07049.x. Epub 2012 Feb 11. PMID 22324297
- [Background] Collins SR, Blank RS. Fiberoptic intubation: an overview and update. Respir Care. 2014 Jun;59(6):865-78; discussion 878-80. doi: 10.4187/respcare.03012. PMID 24891196
- [Background] Moore A, Schricker T. Awake videolaryngoscopy versus fiberoptic bronchoscopy. Curr Opin Anaesthesiol. 2019 Dec;32(6):764-768. doi: 10.1097/ACO.0000000000000771. PMID 31356364
- [Background] Tighe PJ, Badiyan SJ, Luria I, Lampotang S, Parekattil S. Robot-assisted airway support: a simulated case. Anesth Analg. 2010 Oct;111(4):929-31. doi: 10.1213/ANE.0b013e3181ef73ec. PMID 20870983
- [Background] Hemmerling TM, Wehbe M, Zaouter C, Taddei R, Morse J. The Kepler intubation system. Anesth Analg. 2012 Mar;114(3):590-4. doi: 10.1213/ANE.0b013e3182410cbf. Epub 2011 Dec 20. PMID 22190550
- [Background] Hemmerling TM, Taddei R, Wehbe M, Zaouter C, Cyr S, Morse J. First robotic tracheal intubations in humans using the Kepler intubation system. Br J Anaesth. 2012 Jun;108(6):1011-6. doi: 10.1093/bja/aes034. Epub 2012 Mar 28. PMID 22457483
- [Background] Favretto DO, Silveira RC, Canini SR, Garbin LM, Martins FT, Dalri MC. Endotracheal suction in intubated critically ill adult patients undergoing mechanical ventilation: a systematic review. Rev Lat Am Enfermagem. 2012 Sep-Oct;20(5):997-1007. doi: 10.1590/s0104-11692012000500023. English, Portuguese, Spanish. PMID 23174846
- [Background] Haghighat S, Yazdannik A. The practice of intensive care nurses using the closed suctioning system: An observational study. Iran J Nurs Midwifery Res. 2015 Sep-Oct;20(5):619-25. doi: 10.4103/1735-9066.164509. PMID 26457102